CLINICAL TRIAL: NCT04536220
Title: Establish a Diagnostic Model Based on Multiple Molecule Profiling and Certain Established Markers for Identification of Pancreatic Cancer
Brief Title: Establish Diagnostic Models Based on Portal Venous Blood for Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Prefessor of Department of Gastroenterology, Changhai Hospital
Other Study IDs: EMPVC
Record Dates: First submitted 2020-08-18; First posted 2020-09-02 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Diagnoses Disease
Keywords: diagnosis and pancreatic cancer
MeSH Terms: conditions — Disease; Pancreatic Neoplasms | interventions — Endosonography; Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimen collected from pancreatic mass through EUS-FNA, blood collected from portal vein through EUS-FNA, as well as peripheral blood from the patients with pancreatic mass suspicious of malignant pancreatic tumor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pancreatic mass diagnosed benign: Through pathological examination, radiological examination and follow-up, these patients are finally diagnosed with benign pancreatic mass.
  Interventions: Diagnostic Test: Endoscopic Ultrasound (EUS), Fine Needle Aspiration
- pancreatic mass diagnosed malignant: Through pathological examination, radiological examination and follow-up, these patients are finally diagnosed with pancreaitic cancer.
  Interventions: Diagnostic Test: Endoscopic Ultrasound (EUS), Fine Needle Aspiration

INTERVENTIONS:
Diagnostic Test: Endoscopic Ultrasound (EUS), Fine Needle Aspiration — Endoscopic Ultrasound (EUS), Fine Needle Aspiration, which are routine clinical operations

SUMMARY:
Explore new markers based on portal venous blood sampling to establish novel diagnostic models for identification of malignant pancreatic mass.

DETAILED DESCRIPTION:
EUS-FNA combined cytology detection is an important method for clinical diagnosis of squamous cell carcinoma. However, due to factors such as sampling method, smear making, staining technique, lower levels of the pathologists and other factors, its diagnostic sensitivity is still not very satisfactory. Poor diagnostic efficacy usually means another puncture, longer hospital stay, more medications and a higher incidence of adverse events. Missed diagnosis continuously directly delays the treatment time of the disease and seriously affects the patient's prognosis. Therefore, how to use new technologies to improve the differential diagnosis efficiency of benign and malignant pancreatic occupants is the key to improving the prognosis of diabetic cancer patients.

The portal vein blood comes from the venous tract, including the blood flowing from the plasma to the liver. By collecting blood samples from the patient's portal vein, clinicians can separate more information from the patient. Studies have shown that the portal vein blood can be collected by ultrasound endoscopic puncture. This method is less traumatic, convenient and safe, and more information about the retinal tissue can be obtained. It is an important way to improve the efficiency of patient diagnosis. This study intends to use ultrasound endoscopic puncture technology to obtain portal vein blood, and use big data and ctDNA, metabolomics, exosomes and other different omics methods to screen the potential value of volume-occupying benign and malignant differential diagnosis markers in portal vein blood. Peripheral blood will simultaneously be collected to evaluate the efficacy of these newly developed markers.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years,male or female
2. diagnosis or suspection of solid pancreatic mass based on previous imaging examination (ultrasonography, CT or MRI)
3. lesion diameter larger than 1 cm
4. signed informed consent letter

Exclusion Criteria:

1. pregnant female
2. Pancreatic cystic lesions
3. Anticoagulant/antiplatelet therapy cannot be suspended
4. unable or refuse to provide informed consent
5. Coagulopathy (platelet count < 50× 103/μL,international normalized ratio > 1.5)
6. Severe cardiopulmonary dysfunction that cannot tolerate intravenous anesthesia
7. with history of mental disease
8. other medical conditions that are not suitable for EUS-FNA

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion criteria, but not the exclusion criteria, will be included in current study. Pancreatic mass tissue samples, portal venous blood, and periferal blood will be collected for identification of potential markers for diagnosis of malignant pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Status of survival | through study completion, an average of 1 year
  To varify if the patients died becaused of malignant pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Kaixuan Wang, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Within six months this study has been finished